CLINICAL TRIAL: NCT02843763
Title: Study of Specific CD4 Tumors Th1 Responses in Renal Transplant After Occurrence of Cancer
Acronym: TRAK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: University Hospital, Lille (Other); University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: API/2015/59
Record Dates: First submitted 2016-07-19; First posted 2016-07-26 (Estimated); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Disorder Related to Renal Transplantation; Cancer
MeSH Terms: conditions — Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Renal transplant with 1rst cancer (Other): Renal transplant patients with first cancer (all cancer excepting skin cancer including in group 2).
  Intervention : blood sample
  Interventions: Other: Blood sample
- Renal transplant patients without cancer (Other): Renal transplant patients without cancer matched for age, transplantation duration and CMV/EBV status.
  Intervention : blood sample
  Interventions: Other: Blood sample
- Patient with cancer (No Intervention): Patient with cancer from oncology departement matched for cancer type and stade and CMV/EBV status.
- Renal transplant with first skin cancer (Other): Renal transplant patients with first epidermoid skin cancer. Intervention : blood sample
  Interventions: Other: Blood sample
- RT with several skin cancer (Other): Renal transplant patients with several epidermoid skin cancer. Intervention : blood sample
  Interventions: Other: Blood sample
- Rt patients without cancer apparied to RT skin cancer (Other): Renal transplant patients without cancer matched for age, transplantation duration and CMV/EBV status with renal transplant patients with skin cancer.
  Intervention : blood sample
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — Blood sample (28 ml)
  Arms: RT with several skin cancer; Renal transplant patients without cancer; Renal transplant with 1rst cancer; Renal transplant with first skin cancer; Rt patients without cancer apparied to RT skin cancer

SUMMARY:
As early complications of transplantation (acute rejection and infections) were better controlled and that the survival of kidney transplants has increased, chronic complications of immunosuppression became increasing challenges. The incidence of cancer is greatly increased in transplant and cancer is now the first cause of death. The iatrogenic immunosuppression plays a major role in the increased incidence of cancer. If it is accepted that the incidence of cancer is generally increased after transplantation, the increased risk is very different from a specific cancer to another. Furthermore the specific treatment of the tumor (surgery, radiotherapy, chemotherapy, biotherapy), the specificity of the context of transplantation is related to the possibility of modulation of immunosuppression. However, there is no immunological marker for predicting the effectiveness of a modification of the immunosuppression.

Several studies point to the important role of CD4 T cells into Th1 anti-tumor immunosurveillance group cancers. Identified "helper" degenerate peptides, called Universal Cancer Peptide (UCP) derivative of telomerase, a type of tumor antigen universal. These UCP peptides bind most HLA-DR alleles most frequent of the population and have the particularity of specifically stimulate CD4 T cells of type Th1. Using a test based on the UCP, it possible to detect the presence of spontaneous CD4 Th1 anti-UCP answers in several types of human cancers.

The main objective of this study is to determine whether, in renal transplant patients, the occurrence of cancer is associated with a deficiency of CD4 Th1 response anti-hTERT.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 to 80 years included
* Signature of informed consent for participation indicating that the subject has understood the purpose and procedures required by the study and agrees to participate in the study and comply with the requirements and limitations inherent in this study
* Join a French social security or receiving such a plan
* Group 1A: renal transplant patients reporting a first cancer (all types of cancer except skin inclued in group 2A or 2B)
* Group 1B: renal transplant patients without cancer (matched to patients in group 1A)
* 1C Group: Non transplant patients reporting a first cancer (patients matched to Group 1A for the type and stage of cancer and the status CMV / EBV)
* Group 2A: kidney transplant patients reporting a single squamous cell carcinoma
* Group 2B: kidney transplant patients with multiple recurrences of squamous cell carcinomas.
* Group 2C: renal transplant patients without cancer (matched to patients in group 2A and 2B)

Exclusion Criteria:

* Legal incapacity or limited legal capacity
* Topic unlikely to cooperate in the study and / or low early cooperation by the investigator
* Without health insurance Topic
* Pregnant woman
* Inability to understand the reasons for the study; psychiatric disorders judged by the investigator to be incompatible with the inclusion in the study
* Active infection or not by HIV

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2016-07-13 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Th1 anti-hTERT cell serum levels 1A and 1B group | 1 day
  Th1 anti-hTERT cell levels measured in blood by IFN-γ ELISpot in renal transplant patients developing cancer versus first with renal transplant patients without cancer.

SECONDARY OUTCOMES:
Th1 anti-hTERT cell serum levels 1C, 2A and 2B group | 1 day
  Th1anti-hTERT cell levels measured in blood by IFN-γ ELISpot in patients developing a first or recurrent squamous cell carcinoma compared with renal transplant patients without cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Didier Ducloux, Pr., Principal Investigator — Besancon University Hospital, Nephrology department
Locations (1):
- Besançon University Hospital, Besançon, France

IPD SHARING:
Plan to Share IPD: No